CLINICAL TRIAL: NCT04409886
Title: The Application of Hyperbaric Oxygen Therapy in Non-ventilated COVID-19 Patients - Randomized Controlled Trial
Brief Title: Hyperbaric Oxygen Therapy in Non-ventilated COVID-19 Patients
Acronym: HBOT
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: This study is part of a larger national study. Only 1 patient was enrolled at Maimonides; Medical Center. The study was ended by the sponsor because the PI left; funding ended; , and no time, or personnel to do the study
Sponsor: Maimonides Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 120-20-ASF
Record Dates: First submitted 2020-05-27; First posted 2020-06-01 (Actual); Results first posted 2021-06-29 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: COVID, Coronavirus
MeSH Terms: conditions — Coronavirus Infections | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- HBOT (Hyperbaric Oxygen Therapy) (Experimental): Hyperbaric Oxygen Therapy in Non-ventilated COVID-19 Patients (HBOT)
  Interventions: Biological: Hyperbaric Oxygen Therapy

INTERVENTIONS:
Biological: Hyperbaric Oxygen Therapy — Hyperbaric Oxygen Therapy in Non-ventilated COVID-19 Patients (HBOT)

SUMMARY:
This study is a prospective randomized controlled, double blind clinical trial performed on laboratory confirmed COVID-19 infection admitted patients in the Shamir Medical Center. The trial will include 30 patients who will undergo either hyperbaric oxygen therapy (HBOT) or Normobaric oxygen therapy (NBOT), randomized on a 2:1 ratio, within 4 days in addition to the standard treatment including oxygen, drugs, steroids, bronchodilators, antibiotics and others.

The evaluation procedure includes symptom monitoring, room air saturation, vital signs monitoring, pulmonary function and blood tests at baseline, one day and one week after the last session. In addition, one hour prior to and post session saturation and vitals will be monitored.

DETAILED DESCRIPTION:
This study is a prospective randomized controlled, double blind clinical trial performed on laboratory confirmed COVID-19 infection admitted patients at MMC. The trial will include 30 patients who will undergo either HBOT or NBOT, randomized on a 2:1 ratio, within 4 days in addition to the standard treatment including oxygen, drugs, steroids, bronchodilators, antibiotics and others.

Sessions will be provided in an MMC monoplace HBO chamber (RestorixHealth). Since all patients demand oxygen supply at room air, the control group is an active arm receiving 100% oxygen. For HBOT, each session will include breathing 100% oxygen at 2.2 absolute atmospheres (ATA) for 60 minutes. Compression and decompression will occur at 1 meter/minute rate. For NBOT, each session will include breathing 100% oxygen at 1.0 absolute atmospheres (ATA) for 60 minutes. In order to blind the patient, the first 5 minutes will include compression for 1.1 ATA and then decompression to 1.0 within the next 5 minutes.

During the sessions, the symptoms and vitals will be monitored. The evaluation procedure will include symptom monitoring, room air saturation, vital signs monitoring, pulmonary function and blood tests at baseline, one day and one week after the last session. In addition, one hour prior to and post session saturation and vitals will be monitored. Sessions and evaluations procedures will occur as the following:

Protocol Day 1

1. Baseline evaluation: blood test including: arterial blood gases, 2 CBC tubes, 2 Gel tubes (10-15 cc total), vitals (temperature, blood pressure, heart rate, room air saturation), symptoms questionnaire, pulmonary function test.
2. Vitals (temperature, blood pressure, heartrate, room air saturation) one hour prior to session
3. One-hour session NBO/HBO
4. Vitals (temperature, blood pressure, heartrate, room air saturation) one hour after the session.
5. Vitals (temperature, blood pressure, heartrate, room air saturation) one hour before the 2nd session.
6. One-hour session NBO/HBO (8 hours following the first session)
7. Vitals (temperature, blood pressure, heartrate, room air saturation) one hour after the session.
8. Daily oxygen supply dose monitoring. Protocol Day 2-4

1. Daily symptoms questionnaire 2. Vitals (temperature, blood pressure, heartrate, room air saturation) one hour prior to session One-hour session NBO/HBO 3. Vitals (temperature, blood pressure, heartrate, room air saturation) one hour after the session.

4. Vitals (temperature, blood pressure, heartrate, room air saturation) one hour before the 2nd session.

5. One-hour session NBO/HBO (8 hours following the first session) 6. Vitals (temperature, blood pressure, heartrate, room air saturation) one hour after the session.

7. Daily oxygen supply dose monitoring. Follow up Protocol

1. Repeat evaluations one day after the last session and one week after the last session:

   * Blood test including: arterial blood gases, 2 CBC tubes, 2 Gel tubes (10-15 cc total)
   * Vitals (temperature, blood pressure, heart rate, room air saturation)
   * Symptoms questionnaire
   * Pulmonary function test.
2. Oropharyngeal swab for SARS-CoV-2 RT-PCR every 3 days for 1 week
3. Clinical monitoring for 30 days

ELIGIBILITY:
Inclusion Criteria:

* Within 7 days of patient's need of oxygen supply
* Positive SARS-CoV-2 RT-PCR
* At least one risk factor for bad prognosis of COVID-19: hypertension, diabetes mellitus, ischemic heart disease, smoking, age>50, etc.
* Respiratory insufficiency: Room Air SpO2 <94% or PaO2/FiO2<300mmHg
* Age>18
* Ability to sign an informed consent

Exclusion Criteria:

* Negative SARS-CoV-2 RT-PCR
* HBOT contraindication: pneumothorax, pneumomediastinum, claustrophobia, ear/sinus disease which aren't allowed in HBOT, known chronic pulmonary disease: severe emphysema or known pulmonary bullae.
* Pregnancy
* Inability to sign an informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ory Wiesel, MD, Principal Investigator — Maimonides Medical Center
Locations (1):
- Maimonides Medical Center, Brooklyn, New York, United States

IPD SHARING:
Plan to Share IPD: No
Data will not be shared

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | HBOT (Hyperbaric Oxygen Therapy)
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | HBOT (Hyperbaric Oxygen Therapy)
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Oxygenation Index
Description: PaO2/FiO2 (Oxygenation Index)
Time Frame: one day after the last session
Population: PI left institution and the study was terminated with only 1 participant enrolled. No data available to report
Arm/Group | HBOT (Hyperbaric Oxygen Therapy)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 30 days
Description: Adverse events includes adverse events that result in any of the following outcomes: death, a life-threatening adverse event, inpatient hospitalization or prolongation of existing hospitalization, a persistent or significant incapacity or substantial disruption of the ability to conduct normal functions
Arm/Group | HBOT (Hyperbaric Oxygen Therapy)
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-17): https://cdn.clinicaltrials.gov/large-docs/86/NCT04409886/Prot_SAP_000.pdf